CLINICAL TRIAL: NCT02753751
Title: Optimizing Electronic Alerts for Acute Kidney Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1604017596; YALEAKIALERT (Other: former unique ID); 1R01DK113191-01A1 (NIH)
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Results first posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): No alert will be fired.
- Electronic AKI Alert (Experimental): A pop-up alert will fire when a provider opens the electronic health record of a patient with AKI until such time as AKI is documented in the problem list, or AKI resolves.
  Interventions: Other: AKI Alert

INTERVENTIONS:
Other: AKI Alert — Provider's will receive a "pop-up" alert in the electronic health record until AKI is documented in the problem list or AKI resolves.
  Arms: Electronic AKI Alert

SUMMARY:
This study will enroll hospitalized adults with acute kidney injury (AKI) and randomize them to usual care versus an electronic alert coupled to a "best practices" order set.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) carries a significant, independent risk of mortality among hospitalized patients. Recent studies have demonstrated increased mortality among patients with even small increases in serum creatinine concentration. International guidelines for the treatment of AKI focus on appropriate management of drug dosing, avoiding nephrotoxic exposures, and careful attention to fluid and electrolyte balance. Early nephrologist involvement may also improve outcomes in AKI. Without appropriate provider recognition of AKI, however, none of these measures can be taken, and patient outcomes may suffer. AKI is frequently overlooked by clinicians, but carries a substantial cost, morbidity and mortality burden.

The investigators conducted a pilot, randomized trial of electronic alerts for acute kidney injury in 2014. The trial, which randomized 2400 patients with AKI as defined by an increase in creatinine of 0.3mg/dl over 48 hours or 50% over 7 days, found that alerting physicians to the presence of AKI did not improve the course of acute kidney injury, reduce dialysis or death rates. However this study was conducted in a single hospital, and the alert itself did not describe specific actions that a provider could take. In the present proposal, the investigators seek to expand upon their prior study to determine both the modes of alerting that would be most effective and to determine if targeting alerts (such as to patients on medications that may worsen acute kidney injury) will improve effectiveness.

This study will be a randomized, controlled trial of an electronic AKI alert system. Using the Kidney Disease: Improve Global Outcomes creatinine criteria, inpatients at several hospitals will be randomized to usual care versus electronic alerting. The primary outcome will be a composite of progression of acute kidney injury, dialysis and death.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years admitted to a participating study hospital
* Acute Kidney Injury as defined by KDIGO consensus creatinine criteria (0.3mg/dl increase in serum creatinine over 48 hours or 50% relative increase over 7 days).

Exclusion Criteria:

* ESKD diagnosis code
* Dialysis order prior to AKI onset
* Initial creatinine >=4.0mg/dl
* Prior admission in which patient was randomized.
* Admission to hospice service or comfort measures only order
* Kidney transplant within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6030 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis P Wilson, MD MSCE, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified aggregate data for the primary and secondary outcomes will be made available.
Supporting Information: Study Protocol
Time Frame: Data will be available within one year of completion.

REFERENCES:
- [Background] Wilson FP, Shashaty M, Testani J, Aqeel I, Borovskiy Y, Ellenberg SS, Feldman HI, Fernandez H, Gitelman Y, Lin J, Negoianu D, Parikh CR, Reese PP, Urbani R, Fuchs B. Automated, electronic alerts for acute kidney injury: a single-blind, parallel-group, randomised controlled trial. Lancet. 2015 May 16;385(9981):1966-74. doi: 10.1016/S0140-6736(15)60266-5. Epub 2015 Feb 26. PMID 25726515
- [Derived] Wissel BD, Percy Z, Zachem TJ, Beaulieu-Jones B, Kohane IS, Goldstein SL, Gecili E, Dexheimer JW. Heterogenous effect of automated alerts on mortality. J Am Med Inform Assoc. 2025 Dec 25:ocaf222. doi: 10.1093/jamia/ocaf222. Online ahead of print. PMID 41445428
- [Derived] Wissel BD, Percy Z, Zachem TJ, Beaulieu-Jones B, Kohane IS, Goldstein SL, Gecili E, Dexheimer JW. Heterogeneous Effect of Automated Alerts on Mortality. medRxiv [Preprint]. 2025 Aug 13:2025.08.11.25333302. doi: 10.1101/2025.08.11.25333302. PMID 40832403
- [Derived] Wilson FP, Martin M, Yamamoto Y, Partridge C, Moreira E, Arora T, Biswas A, Feldman H, Garg AX, Greenberg JH, Hinchcliff M, Latham S, Li F, Lin H, Mansour SG, Moledina DG, Palevsky PM, Parikh CR, Simonov M, Testani J, Ugwuowo U. Electronic health record alerts for acute kidney injury: multicenter, randomized clinical trial. BMJ. 2021 Jan 18;372:m4786. doi: 10.1136/bmj.m4786. PMID 33461986
- [Derived] Mutter M, Martin M, Yamamoto Y, Biswas A, Etropolski B, Feldman H, Garg A, Gourlie N, Latham S, Lin H, Palevsky PM, Parikh C, Moreira E, Ugwuowo U, Wilson FP. Electronic Alerts for Acute Kidney Injury Amelioration (ELAIA-1): a completely electronic, multicentre, randomised controlled trial: design and rationale. BMJ Open. 2019 Jun 1;9(5):e025117. doi: 10.1136/bmjopen-2018-025117. PMID 31154298
- See also: This link is displayed on the alert and is our clinical trial study website. It contains information about the trial, describes AKI best practices, and provides contact information. — http://akistudy.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 3/29/2018 to 12/14/2019, 6,030 individuals met enrollment criteria and were randomized across 6 hospitals of a single healthcare system.
Period: Overall Study
Arm/Group | Usual Care | Electronic AKI Alert
Started | 2971 | 3059
Completed | 2971 | 3059
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Electronic AKI Alert | Total
Number analyzed (Participants) | 2971 | 3059 | 6030
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71.3 [59.4 to 81.6] | 71 [59 to 81.7] | 71.2 [59.2 to 81.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1440 | 1442 | 2882
  Male | 1531 | 1617 | 3148
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 289 | 331 | 620
  Not Hispanic or Latino | 2664 | 2712 | 5376
  Unknown or Not Reported | 18 | 16 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 8 | 14
  Asian | 35 | 40 | 75
  Native Hawaiian or Other Pacific Islander | 4 | 3 | 7
  Black or African American | 462 | 484 | 946
  White | 2208 | 2234 | 4442
  More than one race | NA — Was not collected. Collected primary race only. | NA — Was not collected. Collected primary race only. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 19 | 23 | 42
Region of Enrollment [Number; unit: participants]
  United States | 2971 | 3059 | 6030
Medical Admission [Count of Participants; unit: Participants] | 2280 | 2284 | 4564
ICU Patient [Count of Participants; unit: Participants] | 961 | 962 | 1923
ER Patient [Count of Participants; unit: Participants] | 108 | 93 | 201
Ward Patient [Count of Participants; unit: Participants] | 1902 | 2004 | 3906
Hospital 1 (Urban, teaching) [Count of Participants; unit: Participants] | 1238 | 1277 | 2515
Hospital 2 (Urban, teaching) [Count of Participants; unit: Participants] | 599 | 649 | 1248
Hospital 3 (Urban, teaching) [Count of Participants; unit: Participants] | 456 | 479 | 935
Hospital 4 (Suburban, teaching) [Count of Participants; unit: Participants] | 292 | 275 | 567
Hospital 5 (Suburban, non-teaching) [Count of Participants; unit: Participants] | 278 | 276 | 554
Hospital 6 (Suburban, non-teaching) [Count of Participants; unit: Participants] | 108 | 103 | 211
Chronic Kidney Disease [Count of Participants; unit: Participants] | 1127 | 1163 | 2290
Congestive Heart Failure [Count of Participants; unit: Participants] | 1307 | 1351 | 2658
COPD [Count of Participants; unit: Participants] | 1015 | 1049 | 2064
Diabetes Mellitus [Count of Participants; unit: Participants] | 1197 | 1287 | 2484
Hypertension [Count of Participants; unit: Participants] | 2434 | 2510 | 4944
Malignancy [Count of Participants; unit: Participants] | 471 | 460 | 931
Depression [Count of Participants; unit: Participants] | 687 | 655 | 1342
Liver Disease [Count of Participants; unit: Participants] | 397 | 458 | 855
eGFR at admission (ml/min/1.73m2) [Median (Inter-Quartile Range); unit: ml/min/1.73m2] | 55.1 [34.2 to 84.4] | 55.8 [36.6 to 83.5] | 55.4 [35.3 to 83.9]
Creatinine, mg/dL [Median (Inter-Quartile Range); unit: mg/dL] | 1.5 [1.1 to 2] | 1.5 [1.2 to 2] | 1.5 [1.2 to 2]
Nadir creatinine in 48 hrs prior to randomization, mg/dL [Median (Inter-Quartile Range); unit: mg/dL] | 1.1 [0.8 to 1.5] | 1.1 [0.8 to 1.5] | 1.1 [0.8 to 1.5]
Sodium, meq/L [Median (Inter-Quartile Range); unit: meq/L] | 138 [135 to 141] | 138 [135 to 141] | 138 [135 to 141]
Potassium, meq/L [Median (Inter-Quartile Range); unit: meq/L] | 4.2 [3.8 to 4.6] | 4.2 [3.8 to 4.6] | 4.2 [3.8 to 4.6]
Chloride, meq/L [Median (Inter-Quartile Range); unit: meq/L] | 102 [98 to 106] | 102 [98 to 106] | 102 [98 to 106]
Bicarbonate, meq/L [Median (Inter-Quartile Range); unit: meq/L] | 24 [21 to 27] | 24 [21 to 27] | 24 [21 to 27]
Anion Gap, meq/L [Median (Inter-Quartile Range); unit: meq/L] | 12 [10 to 14] | 12 [10 to 15] | 12 [10 to 15]
Blood Urea Nitrogen, mg/dL [Median (Inter-Quartile Range); unit: mg/dL] | 28 [18 to 42] | 28 [19 to 40] | 28 [19 to 41]
White Blood Cell Count, (cells*1000/ul) [Median (Inter-Quartile Range); unit: cells*1000/uL] | 9.8 [7.2 to 13.5] | 9.8 [7.2 to 13.8] | 9.8 [7.2 to 13.6]
Hemoglobin, g/dL [Median (Inter-Quartile Range); unit: g/dL] | 10.7 [9 to 12.3] | 10.5 [8.9 to 12.3] | 10.6 [9 to 12.3]
Platelet Count, (cells*1000/ul) [Median (Inter-Quartile Range); unit: cells*1000/ul] | 202.5 [149 to 266] | 200 [144 to 266] | 201 [146 to 266]
Contrast in prior 72 hours [Count of Participants; unit: Participants] | 586 | 623 | 1209
Cardiothoracic surgery in prior 72 hours [Count of Participants; unit: Participants] | 110 | 135 | 245
ACE inhibitor/ARB in prior 72 hours [Count of Participants; unit: Participants] | 626 | 670 | 1296
NSAID in prior 72 hours [Count of Participants; unit: Participants] | 403 | 388 | 791
PPI in prior 72 hours [Count of Participants; unit: Participants] | 684 | 677 | 1361
Time from admission to randomization, hours [Median (Inter-Quartile Range); unit: hours] | 50.7 [28.8 to 104.3] | 50.1 [29.8 to 101.0] | 50.3 [29.3 to 103.2]
Time from AKI to randomization, hours [Median (Inter-Quartile Range); unit: hours] | 0.5 [0.2 to 1.3] | 0.5 [0.2 to 1.2] | 0.5 [0.2 to 1.3]
Unique providers reached [Median (Inter-Quartile Range); unit: Providers] | 7 [4 to 13] | 7 [4 to 13] | 7 [4 to 13]

OUTCOME MEASURES:

1. Primary Outcome: Composite of Progression of AKI, Inpatient Dialysis, or Inpatient Death
Description: Progression of AKI is defined by an increase in KDIGO creatinine stage from that present at the time of randomization.
  Dialysis is defined by the receipt of hemodialysis, continuous renal replacement therapy or peritoneal dialysis. Isolated ultrafiltration treatments (for the purpose of volume removal) will not be included.
  Mortality will be determined from hospital administrative records.
Time Frame: 14 days from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Electronic AKI Alert
Number analyzed (Participants) | 2971 | 3059
Participants | 622 | 653
Statistical Analysis 1: Comparison: Usual Care vs Electronic AKI Alert; In our retrospective analysis of patients with AKI at 3 potential study hospitals, the composite outcome was 24.5%. A clinically meaningful relative reduction in this risk would be 20%. 5,024 patients (2,512 in each group) would have 90% power to detect a difference in outcome at least this extreme at a two-sided alpha of 0.05 as calculated using the Cochran-Mantel-Haenszel test. We have elected to increase this number by 20% to account for potential contamination; Test type: Superiority — The Mantel-Haenszel test was used, accounting for each hospital as an individual stratum, and to obtain the pooled relative risks across hospitals without adjusting for other baseline factors. (Alert arm is the numerator, control arm is the denominator.) Patients discharged prior to 14 days without an outcome of interest were assumed to be free of that outcome at 14 days. A p-value of <=0.04 was considered statistically significant to account for the interim analysis; p = 0.67, Cochran-Mantel-Haenszel — A p-value of <=0.04 was considered statistically significant to account for the interim analysis; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.93 to 1.13]

2. Secondary Outcome: Mortality
Description: 14-day or inpatient mortality
Time Frame: 14 days from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Electronic AKI Alert
Number analyzed (Participants) | 2971 | 3059
Participants | 265 | 272

3. Secondary Outcome: Dialysis
Description: 14-day, inpatient, or discharged on dialysis
Time Frame: 14 days from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Electronic AKI Alert
Number analyzed (Participants) | 2971 | 3059
Participants | 93 | 106

4. Secondary Outcome: AKI Progression
Description: Percent of patients who progress to stage 2 AKI and to stage 3 AKI
Time Frame: 14 days from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Electronic AKI Alert
Number analyzed (Participants) | 2971 | 3059
Participants | 461 | 487

5. Secondary Outcome: AKI Duration
Description: Number of participants with AKI duration of <2 days, 2-<days, and 7+ days (Aki duration defined as time in days between AKI onset and AKI cessation during index hospitalization)
Time Frame: 14 days from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Electronic AKI Alert
Number analyzed (Participants) | 2971 | 3059
Participants
  <2 days | 2108 | 2239
  2-<7 days | 722 | 700
  7+ days | 141 | 120

6. Secondary Outcome: Readmission Rate
Description: 30 day readmission rate
Time Frame: 30 days from randomization
Population: Data have not yet been collected.
Arm/Group | Usual Care | Electronic AKI Alert
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Index Hospitalization Cost
Description: Cost of index hospitalization, measured in direct and total costs. Direct costs reflect those associated with direct patient contact involving billable services (for example lab, nursing costs, and supplies). Total costs also include non-billable support services such as medical records, human resources, accounting, support staff, utilities and dietary costs.
Time Frame: Index hospitalization through discharge, up to one year
Measure: Median (Inter-Quartile Range); unit: dollars
Arm/Group | Usual Care | Electronic AKI Alert
Number analyzed (Participants) | 2971 | 3059
dollars
  Direct Costs | 10300 [5400 to 21900] | 10600 [5400 to 22800]
  Total Costs | 19100 [9900 to 42500] | 20100 [10200 to 43600]

8. Secondary Outcome: Proportion of AKI "Best Practices" Achieved Per Subject During Index Hospitalization
Description: Best practices assessed include: Avoidance of nephrotoxins (cessation of order or absence of de novo order of IV contrast agent, aminoglycoside, NSAID, or ACE inhibitor within 24 hours of randomization), fluid administration (administration of fluids within 24 hours of randomization), urinalysis order (with or without microscopy within 24 hours of randomization), documentation of AKI (by ICD-9 and ICD-10 codes during index hospitalization), monitoring of creatinine (at least one serum creatinine measurement occurring within 36 hours of randomization), documentation of urine output (within 24 hours of randomization), renal consult order during index hospitalization.
  Each metric above is binary. Outcome is reported as a composite best practice outcome representing the proportion of best practices achieved per subject.
Time Frame: 24 hours from randomization to discharge, up to one year
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Electronic AKI Alert
Number analyzed (Participants) | 2971 | 3059
Participants
  IV fluid drip order | 1034 | 1174
  IV fluid bolus order | 339 | 397
  Urinalysis | 444 | 519
  Urine Output Measurement | 2130 | 2242
  Subsequent Creatinine Measurement (28 hours) | 2532 | 2666
  Renal Consult (within 14 days) | 517 | 541
  Contrast exposure | 102 | 115
  Aminoglycoside exposure | 19 | 14
  Aminoglycoside exposure among those already receiving aminoglycoside | 8 | 5
  NSAID exposure | 166 | 144
  NSAID exposure among those already receiving NSAIDs | 129 | 103
  ACE/ARB exposure | 425 | 424
  ACE/ARB exposure among those already receiving ACE/ARB | 326 | 331
  AKI documentation (at end of encounter) | 1871 | 2141

9. Secondary Outcome: Number of Subjects With Chart Documentation of AKI
Description: Proportion of subjects with chart documentation of AKI by post-discharge ICD-10 codes and by chart adjudication
Time Frame: Index hospitalization
Population: Chart documentation via ICD-10 codes (code N17) have been collected. Documentation via chart adjudication has not yet been collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Electronic AKI Alert
Number analyzed (Participants) | 2971 | 3059
Participants | 1871 | 2141

ADVERSE EVENTS:
Time Frame: Duration of the study (22 months)
Arm/Group | Usual Care | Electronic AKI Alert
All-Cause Mortality (participants affected / at risk) | 265/2971 | 272/3059
Serious Adverse Events (participants affected / at risk) | 0/2971 | 0/3059
Other Adverse Events (participants affected / at risk) | 0/2971 | 0/3059

LIMITATIONS AND CAVEATS:
Randomization occurred at the patient level, potentially biasing the results towards the null hypothesis.

The alert was largely informational with no patient-specific recommendations.

The alert was only sent to certain care providers, notably excluding nurses and pharmacists, who might specifically benefit from receipt of the alert.

The alert was conducted across six hospitals within a single large health system in the Northeastern United States, limiting generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT02753751/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT02753751/SAP_001.pdf